CLINICAL TRIAL: NCT03796962
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Safety, Tolerability and Efficacy of XEN1101 as Adjunctive Therapy in Focal-onset Epilepsy, With an Open-label Extension
Brief Title: A Study to Evaluate XEN1101 as Adjunctive Therapy in Focal Epilepsy
Acronym: X-TOLE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Collaborators: Novotech Health Holdings Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XPF-008-201; 2018-003221-29 (EudraCT Number)
Record Dates: First submitted 2019-01-02; First posted 2019-01-08 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Focal Epilepsy
Keywords: Epilepsy
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — XEN1101

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 25 mg XEN1101 (Experimental): Capsule filled with 25 mg XEN1101
  Interventions: Drug: XEN1101
- 20 mg XEN1101 (Experimental): Capsule filled with 20 mg XEN1101
  Interventions: Drug: XEN1101
- 10 mg XEN1101 (Experimental): Capsule filled with 10 mg XEN1101
  Interventions: Drug: XEN1101
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Drug: XEN1101

INTERVENTIONS:
Drug: XEN1101 — Oral dose

SUMMARY:
The XEN1101 Phase 2 clinical trial is a randomized, double-blind, placebo-controlled study that will evaluate the clinical efficacy, safety and tolerability of increasing doses of XEN1101 administered as adjunctive treatment in adult patients diagnosed with focal epilepsy, followed by an optional open-label extension (OLE).

DETAILED DESCRIPTION:
The XEN1101 Phase 2 clinical trial is designed as a randomized, double-blind, placebo-controlled, multicenter study with an optional open-label extension (OLE) to evaluate the clinical efficacy, safety and tolerability of XEN1101 administered as adjunctive treatment in adult patients aged 18 to 75 years diagnosed with focal epilepsy. Approximately 300 patients will be randomized in a blinded manner to one of three active treatment groups or placebo in a 2:1:1:2 fashion (XEN1101 25 mg : 20 mg : 10 mg : Placebo). After screening, patients will have 8 weeks of baseline to assess frequency of seizures, followed by 8 weeks of treatment and a 6-week post treatment follow-up period. In order to be included in the study, patients must already be treated with a stable dose of 1 to 3 allowable current anti-epileptic drugs for at least one month prior to screening, during baseline, and throughout the double-blind portion (DBP) of the study. During the treatment period, patients will be given XEN1101 or placebo once daily in the evening. An OLE will be available to eligible patients who complete the DBP. All patients will receive a 20 mg daily dose of XEN1101 during this extension period.

ELIGIBILITY:
Key Inclusion Criteria:

* Be properly informed of the nature and risks of the study and give informed consent in writing, prior to entering the study
* BMI ≤40 kg/m2
* Diagnosis (≥2 years) of focal epilepsy according to the International League Against Epilepsy [ILAE] Classification of Epilepsy (2017)
* Prior neuroimaging within the last 10 years and documentation is available
* Treatment with a stable dose of 1 to 3 allowable current AEDs for at least one month prior to screening, during baseline, and throughout the duration of the DBP
* Must be willing to comply with the contraception requirements
* Males must agree not to donate sperm from the time of the first administration of study drug until 6 months after the last dose. Females must agree not to donate ova from the time of the first administration of study drug until 6 months after the last dose.
* Able to keep accurate seizure diaries

Key Exclusion Criteria:

* History of pseudoseizures, psychogenic seizures, primary generalized seizure, or focal aware non-motor seizures only
* Presence or previous history of Lennox-Gastaut syndrome
* Seizures secondary to other diseases or conditions
* History of repetitive seizures within the last 12 months where the individual seizures cannot be counted
* History of neurosurgery for seizures <1 year prior to enrollment, or radiosurgery <2 years prior to enrollment
* Schizophrenia and other psychotic disorders, or active suicidal plan/intent in the past 6 months, or a history of suicide attempt in the last 2 years, or more than 1 lifetime suicide attempt
* History or presence of any significant medical or surgical condition or uncontrolled medical illness at screening, or history of cancer within the past 2 years, with the exception of appropriately treated basal cell or squamous cell carcinoma
* Any clinically significant abnormalities on pre-study physical examination, vital signs, laboratory values or ECG indicating a medical problem that would preclude study participation including but not limited to:

  1. History of presence of long QT syndrome; QTcF > 450 msec at baseline; family history of sudden death of unknown cause
  2. History of skin or retinal pigment epithelium abnormalities caused by ezogabine
* Past use of vigabatrin without stable visual fields tested twice over the 12 months after the last dose of vigabatrin (concomitant use of vigabatrin is not allowed)
* If felbamate is used as a concomitant AED, patients must be taking it for at least 2 years, with a stable dose for 2 months (or no less than 49 days) and acceptable hematology and LFT history and values prior to Screening. If received in the past, felbamate must have been discontinued 2 months (or no less than 49 days) prior to Screening.
* Have had multiple drug allergies or a severe drug reaction to an AED(s), including dermatological (e.g., Stevens-Johnson syndrome), hematological, or organ toxicity reactions
* Current use of a ketogenic diet

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2028-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Xenon Pharmaceuticals Inc.
Locations (95):
- United States (54):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Strada Patient Care Center, Mobile, Alabama
  - Xenoscience, Inc., Phoenix, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - Altman Clinical Translational Research Institute (ACTRI), La Jolla, California
  - California Pacific Medical Center (CPMC) - Sutter Pacific Epilepsy Program, San Francisco, California
  - University of Colorado Hospital Anschutz Outpatient Pavilion, Aurora, Colorado
  - University of Florida Jacksonville, Jacksonville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Visionary Investigators Network, Miami, Florida
  - Don Clinical Research Center, Miami, Florida
  - The Neurology Research Group, LLC., Miami, Florida
  - Research Institute of Orlando, LLC, Orlando, Florida
  - Medsol Clinical Research Center, Port Charlotte, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - University of South Florida, Tampa, Florida
  - Georgia Neurology and Sleep Medicine Associate, Suwanee, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Consultants in Epilepsy and Neurology, PLLC, Boise, Idaho
  - Northwestern Medical Group, Department of Neurology, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Bluegrass Epilepsy Research, Lexington, Kentucky
  - Maine Medical Partners Neurology, Scarborough, Maine
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Boston Neuro Research Center, South Dartmouth, Massachusetts
  - Minneapolis Clinic of Neurology, Ltd., Golden Valley, Minnesota
  - Minnesota Epilepsy Group, P. A., Saint Paul, Minnesota
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Institute of Neurology and Neurosurgery at Saint Barnabas, Livingston, New Jersey
  - Northeast Regional Epilepsy Group, Morristown, New Jersey
  - Dent Neurosciences Research Center, Amherst, New York
  - NYU Langone Medical Center/NYU School of Medicine, New York, New York
  - Northwell Health - Lenox Hill, New York, New York
  - SUNY Upstate Medical University Institute for Human Performance, Syracuse, New York
  - Five Towns Neuroscience Research, Woodmere, New York
  - Asheville Neurology Specialists, PA, Asheville, North Carolina
  - UC Gardner Neuroscience Institute, Cincinnati, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Providence Neurological Specialties East, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Comprehensive Epilepsy Center, Philadelphia, Pennsylvania
  - Allegheny Neurological Associates, Pittsburgh, Pennsylvania
  - Vanderbilt Epilepsy Clinic, Nashville, Tennessee
  - Austin Epilepsy Care Center, Austin, Texas
  - James W. Aston Ambulatory Care Center, Dallas, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah Health Clinical Neurosciences Center, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Carilion Neurology Clinic, Roanoke, Virginia
  - Winchester Neurological Consultants, Winchester, Virginia
  - UW Medicine Valle Medical Center, Renton, Washington
  - University of Washington School of Medicine, Regional Epilepsy Center at Harborview Medical Center, Seattle, Washington
- Canada (3):
  - Children's and Women's Health Centre of British Columbia (BC Children's Hospital), Vancouver, British Columbia
  - London Health Sciences Center, London, Ontario
  - University Health Network-Toronto Western Hospital, Toronto, Ontario
- LLC Arensia Exploratory Medicine, Tbilisi, Georgia
- Germany (9):
  - Epilepsiezentrum Berlin-Brandenburg, Berlin
  - Bethel Epilepsy Centre, Bielefeld
  - Univ.-Klinik Bonn, Klinik und Poliklinik fur Epileptologie, Bonn
  - Universitatsklinikym Frankfurt, Frankfurt
  - Universitatsklinikum Freiburg, Neurozentrum/Epilepsiezentrum, Freiburg im Breisgau
  - University Hospital Munster (UKM), Münster
  - Klinikum Osnabruck, Osnabrück
  - Krankenhaus Barmherzige Brueder Regensburg, Regensburg
  - University of Tubingen-Dept. of Neurology and Epileptology, Tübingen
- Italy (7):
  - IRCCS- Istituto delle Scienze Neurologiche, Bellaria Hospital, Bologna
  - Dipartimento Scienze Mediche e Chirurgiche, Universita Magna Graecia di Catanzaro, Catanzaro
  - Fondazione IRCCS Istituto Neurologico C. Besta, Milan
  - IRCCS Istituto Neurologico Nazionale C. Mondino, Pavia
  - Azienda Ospedaliera Universita' Pisana, Pisa
  - Azienda Ospedaliera "Bianchi-Melacrino-Morelle"di Reggio Calabria, Reggio Calabria
  - Policlinico di Roma Umberto I, Roma
- PMSI Republican Clinical Hospital, ARENSIA Exploratory Medicine, Chisinau, Moldova
- Spain (15):
  - Hospital Virgen Macarena, Seville, Andalusia
  - Centro de Neurologia Avanzada, Seville, Andalusia
  - Hospital Germans Trias I Pujol, Badalona, Barcelona
  - Clínica Universidad Navarra, Pamplona, Navarre
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Vithas La Salud, Granada
  - Hospital U. Ramón y Cajal, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital U. Clínico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Clínico Universitario Valladolid, Valladolid
- Medical Center of Limited Liability Company "Harmoniya Krasy", Kyiv, Ukraine
- United Kingdom (4):
  - Institute of Neurological Sciences, Glasgow, Scotland
  - University Hospital of Wales, Cardiff, Wales
  - King's College Hospital NHS Foundation Trust, London
  - St. George's University Hospitals NHS Foundation Trust, London

REFERENCES:
- [Result] French JA, Porter RJ, Perucca E, Brodie MJ, Rogawski MA, Pimstone S, Aycardi E, Harden C, Qian J, Rosenblut CL, Kenney C, Beatch GN; X-TOLE Study Group. Efficacy and Safety of XEN1101, a Novel Potassium Channel Opener, in Adults With Focal Epilepsy: A Phase 2b Randomized Clinical Trial. JAMA Neurol. 2023 Nov 1;80(11):1145-1154. doi: 10.1001/jamaneurol.2023.3542. PMID 37812429

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 530 subjects were screened; 77 subjects screen failed; 124 subjects that entered the baseline period but were not randomized due seizure/eDiary-based eligibility criteria
Period: Overall Study
Arm/Group | 25 mg XEN1101 | 20 mg XEN1101 | 10 mg XEN1101 | Placebo
Started | 114 | 51 | 46 | 114
Completed | 88 | 43 | 45 | 109
Not Completed | 26 | 8 | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 25 mg XEN1101 | 20 mg XEN1101 | 10 mg XEN1101 | Placebo | Total
Number analyzed (Participants) | 114 | 51 | 46 | 114 | 325
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 38.7 (13.1) | 41.7 (13.6) | 40.0 (12.1) | 42.9 (13.7) | 40.8 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 26 | 27 | 61 | 168
  Male | 60 | 25 | 19 | 53 | 157
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1 | 2 | 4
  Black or African American | 2 | 1 | 2 | 7 | 12
  Native Hawaiian or Other | 1 | 1 | 0 | 1 | 3
  White or Caucasian | 105 | 49 | 42 | 102 | 298
  Other | 5 | 0 | 1 | 2 | 8
Monthly seizure frequency in baseline [Median (Inter-Quartile Range); unit: seizures/month (28 days)] | 12.8 [8.4 to 24.6] | 14.5 [7.5 to 36.4] | 17.4 [8.0 to 55.6] | 13.4 [8.0 to 30.1] | 13.5 [7.9 to 30.3]

OUTCOME MEASURES:

1. Primary Outcome: Median Percent Change in Focal Seizure Frequency
Description: Median percent change in monthly (28 days) focal seizure frequency from baseline to DBP for XEN1101 versus placebo
Time Frame: From baseline (8 weeks prior to Day 0) through to the final dose (up to Day 56)
Population: mITT
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | 25 mg XEN1101 | 20 mg XEN1101 | 10 mg XEN1101 | Placebo
Number analyzed (Participants) | 112 | 51 | 46 | 114
Percent change | -52.8 [-80.4 to -16.9] | -46.4 [-76.7 to -14.0] | -33.2 [-61.8 to 0.0] | -18.2 [-37.3 to 7.0]

2. Secondary Outcome: 50% XEN1101 Response Rate
Description: Responders are defined as patients experiencing ≥50% reduction in monthly (28 days) focal seizure frequency from baseline to DBP
Time Frame: From baseline (8 weeks prior to Day 0) through to the final dose (up to Day 56)
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | 25 mg XEN1101 | 20 mg XEN1101 | 10 mg XEN1101 | Placebo
Number analyzed (Participants) | 112 | 51 | 46 | 114
Participants | 61 | 22 | 13 | 17

3. Secondary Outcome: Percent Change in Focal Seizure Frequency Over Time
Description: Percent change from baseline in focal seizure frequency at Month 1 and Month 2 in the DBP
Time Frame: From baseline (8 weeks prior to Day 0) through to the final dose (up to Day 56)
Population: mITT population
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | 25 mg XEN1101 | 20 mg XEN1101 | 10 mg XEN1101 | Placebo
Number analyzed (Participants) | 112 | 51 | 46 | 114
Percent change from baseline
  Month 1 (Day 1 to 28) | -55.3 [-78.3 to -16.1] | -40.0 [-70.7 to -1.3] | -40.1 [-62.5 to -1.5] | -14.9 [-38.6 to 15.9]
  Month 2 (Day 29 to Visit 8): number analyzed (Participants) | 95 | 45 | 46 | 112
  Month 2 (Day 29 to Visit 8) | -64.7 [-91.1 to -32.8] | -52.2 [-81.1 to -33.7] | -30.3 [-56.9 to 0.3] | -21.8 [-45.6 to 4.9]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | 25 mg XEN1101 | 20 mg XEN1101 | 10 mg XEN1101 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/51 | 0/46 | 0/114
Serious Adverse Events (participants affected / at risk) | 3/114 | 2/51 | 2/46 | 3/114
Other Adverse Events (participants affected / at risk) | 97/114 | 35/51 | 31/46 | 56/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 mg XEN1101 (N=114) | 20 mg XEN1101 (N=51) | 10 mg XEN1101 (N=46) | Placebo (N=114)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychogenic seizure (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somatic delusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasticity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 mg XEN1101 (N=114) | 20 mg XEN1101 (N=51) | 10 mg XEN1101 (N=46) | Placebo (N=114)
Dizziness (Nervous system disorders) | 36 (36) | 13 (13) | 3 (3) | 8 (8)
Somnolence (Nervous system disorders) | 17 (17) | 11 (11) | 5 (5) | 8 (8)
Headache (Nervous system disorders) | 9 (9) | 6 (6) | 6 (6) | 9 (9)
Balance disorder (Nervous system disorders) | 13 (13) | 4 (4) | 2 (2) | 2 (2)
Tremor (Nervous system disorders) | 12 (12) | 3 (3) | 3 (3) | 2 (2)
Aphasia (Nervous system disorders) | 8 (8) | 1 (1) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 5 (5) | 1 (1) | 3 (3) | 1 (1)
Dysarthria (Nervous system disorders) | 8 (8) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 6 (6) | 2 (2) | 1 (1) | 1 (1)
Disturbance in attention (Nervous system disorders) | 5 (5) | 3 (3) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 6 (6) | 3 (3) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 5 (5) | 0 (0) | 6 (6)
Hallucination (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 14 (14) | 4 (4) | 5 (5) | 6 (6)
Gait disturbance (General disorders) | 8 (8) | 2 (2) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7) | 1 (1) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Vision blurred (Eye disorders) | 7 (7) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT03796962/Prot_SAP_001.pdf